CLINICAL TRIAL: NCT04362917
Title: Identification of β Cell Dysfunction in Relatives of Individuals With Type 1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Emily K. Sims, Assistant Professor of Pediatrics, Indiana University
Other Study IDs: T1DFam
Record Dates: First submitted 2020-02-19; First posted 2020-04-27 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- FDR-: Adults with a first degree relative with T1D, who have tested negative for islet autoantibodies.
  There is no intervention. Each group will get a MMTT and a clamp to evaluate beta cell function, identify elevations in circulating biomarkers of β cell stress or death, as well as their associations with measures of β cell function, and compare advantages of hyperglycemic clamps in identifying β cell dysfunction in this setting, relative to the mixed meal tolerance test (MMTT). They will repeat both the MMTT and the clamp once, to assess inter-test variability.
  Interventions: Other: There is no intervention
- FDR+: Adolescents and adults with a first or second degree relative with T1D, who has tested positive for at least one islet autoantibody.
  There is no intervention. Each group will get a MMTT and a clamp to evaluate beta cell function, identify elevations in circulating biomarkers of β cell stress or death, as well as their associations with measures of β cell function, and compare advantages of hyperglycemic clamps in identifying β cell dysfunction in this setting, relative to the mixed meal tolerance test (MMTT). They will repeat both the MMTT and the clamp once, to assess inter-test variability.
  Interventions: Other: There is no intervention
- Control: Adults with no family history of Type 1 Diabetes, who have tested negative for islet autoantibodies
  There is no intervention. Each group will get a MMTT and a clamp to evaluate beta cell function, identify elevations in circulating biomarkers of β cell stress or death, as well as their associations with measures of β cell function, and compare advantages of hyperglycemic clamps in identifying β cell dysfunction in this setting, relative to the mixed meal tolerance test (MMTT). They will repeat both the MMTT and the clamp once, to assess inter-test variability.
  Interventions: Other: There is no intervention

INTERVENTIONS:
Other: There is no intervention — There is no intervention

SUMMARY:
Despite the valuable information derived from older studies evaluating type 1 diabetes, the diabetes research community has, in large part, overlooked potential contributions of baseline abnormalities in β cell function to T1D development. Newer studies focusing on higher risk individuals often exclude family members without evidence of positive islet autoantibodies. New technologies to assay alternative biomarkers of β cell stress and death remain incompletely explored in both Ab negative and Ab positive family members of T1D patients. Specifically, modern biomarkers of β cell dysfunction have not been rigorously tested in combination with metabolic testing to fully understand their association with insulin secretion.

The investigator's working hypothesis is that individuals at genetic risk for T1D exhibit baseline β cell dysfunction, even before development of detectable islet autoimmunity (seropositivity for islet Abs).

ELIGIBILITY:
Inclusion criteria for each subject group* note age limits different for each group*:

* Nonrelative controls: Male and female adults 18-55 years old with no family history of Type 1 Diabetes, who have tested negative for glutamic acid decarboxylase, microinsulin, islet cell, islet antigen 2, and zinc transporter 8 autoantibodies
* Ab negative FDRs: Male and female adults 18-50 years old with a first degree relative (sibling, child, or parent) with T1D, who have tested negative for the above islet autoantibodies
* Ab + T1D Relatives: Male and females aged 12-50 years old with a first or second degree relative diagnosed with T1D, and testing positive for 1 of the above islet autoantibodies either at the screening visit, or through TrialNet screening obtained within the past 12 months.

Criteria for all subjects:

* BMI≤40 kg/m2 (If FDR is 40 kg/m2, the healthy control BMI can not exceed 45 kg/m2)
* HbA1c< 5.7%
* No medical history of diabetes.

Exclusion criteria for all participants:

* Any type of diabetes or hyperglycemia (HbA1c≥5.7%)
* Chronic illness or use of medications which interfere with glucose or islet hormone metabolism.
* Hemoglobin < 12 g/dL
* Presence of any psychiatric disorder that will affect the ability to participate in the study
* Pregnancy
* Severe milk or soy allergy that would disallow Boost® ingestion for MMTT
* Any condition that, in the judgment of the investigator, will adversely affect adequate participation in, or the safety or technical performance of the protocol.

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Comparing a population at risk for T1D to healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Measurement of beta cell function during the first phase of the first clamp procedure | The data for this analysis will come from cross-sectional samples collected through study completion, study completion will be on average 13-16 weeks from visit 1.
  Our primary outcome is to assess if there is a difference in first phase beta call function in those genetically at risk for developing type 1 diabetes (first degree relatives) but who are islet autoantibody negative versus healthy controls with no family history of type 1 diabetes.
  We will calculate the first phase beta cell function by multiplying the acute c-peptide response to glucose (ACPRg) (nmol/L) by the insulin sensitivity (M/I) (x10-5 mmol/kg/min per pmol/L)

SECONDARY OUTCOMES:
Measurement of beta cell function during of Second Phase of the first clamp procedure | The data for this analysis will come from cross-sectional samples collected through study completion, study completion will be on average 13-16 weeks from visit 1.
  Our secondary outcome is to assess if there is a difference in second phase beta cell function in those genetically at risk for developing type 1 diabetes (first degree relatives) but who are islet autoantibody negative versus healthy controls with no family history of type 1 diabetes.
  We will calculate the second phase beta cell function by averaging the C-peptide values collected during the steady state of the clamp (nmol*L) and multiplying by the insulin sensitivity (M/I) (x10-5 mmol/kg/min per pmol/L)

OTHER OUTCOMES:
Measurement of the Unmethylated and methylated DNA as this is a marker of beta cell death | The data for this analysis will come from cross-sectional samples collected through study completion, study completion will be on average 13-16 weeks from visit 1.
  Another prespecified outcome measure is to see if there is a difference in unmethylated/methylated INS DNA (which is a biomarker of beta cell death) in those genetically at risk for developing type 1 diabetes (first degree relatives) but who are islet autoantibody negative versus healthy controls with no family history of type 1 diabetes.
Measurement of the Fasting Proinsulin to the C-peptide ratio (PI:C) | The data for this analysis will come from cross-sectional samples collected through study completion, study completion will be on average 13-16 weeks from visit 1.
  Another prespecified outcome measure is to see if there is a difference in the Proinsulin/C-peptide ratio (PI:C) in those genetically at risk for developing type 1 diabetes (first degree relatives) but who are islet autoantibody negative versus healthy controls with no family history of type 1 diabetes.
Test-retest variability of the above mentioned variables (first phase, second phase, Unmethylated and methylated DNA, fasting PI:C | The data for this analysis will come from cross-sectional samples collected through study completion, study completion will be on average 13-16 weeks from visit 1.
  We will calculate the test-retest variability of the above mentioned variables (first phase, second phase, unmethylated/methylated DNA, fasting proinsulin/c-peptide), by looking at the between-visit coefficients of variation and intraclass correlations.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Sims, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No